

# Official Title: Comparison of Rainbow INVSENSOR00001 and Control SpHb Disposable Sensor Performance during Hemodilution

Date of Protocol: May 8, 2018

NCT Number: NCT03273166

R-TP - 18788

# Comparison of Rainbow INVSENSOR00001 and Control SpHb Disposable Sensor Performance during Hemodilution

| Protocol/Test Procedure Title | Comparison of Rainbow INVSENSOR00001 and Control SpHb Disposable Sensor Performance during Hemodilution |
|---|---|
| Lead Investigator | Tala Harake, MS, BS Senior Clinical Lab Manager Masimo Corporation 52 Discovery, Irvine, CA 92618 |
| Other Investigators | Assistant Clinical lab Manager Masimo Corporation 52 Discovery, Irvine, CA 92618 Clinical Research Associate Masimo Corporation 52 Discovery, Irvine, CA 92618 |
| Expected Start Date | |
| Expected End Date | |
| IRB | E&I West Coast Board – IRB00007807 |
| Protocol Version Date | TBD |

#### **Protocol Test Abstract:**

This study involves comparison of the performance of two SpHb sensors in subjects that undergo a hemodilution procedure. The sensors performance will be assessed by comparison of the measured hemoglobin values against reference values obtained by a laboratory hematology analyzer. Blood samples will be collected from healthy volunteers who undergo a hemodilution procedure wherein blood is repeatedly sampled as the concentration of hemoglobin is reduced by administering intravenous fluids to the volunteer in a controlled manner.

#### **APPROVALS**

| Author | Date | Engineering | Date |
|-------------------|------|---------------|------|
| Quality Assurance | Date | Manufacturing | Date |



R-TP - 18788

Comparison of Rainbow INVSENSOR00001 and Control SpHb Disposable Sensor Performance during Hemodilution

#### STATEMENT OF COMPLIANCE

This document is a protocol for a clinical research study sponsored by Masimo Corporation. The study will be conducted in compliance with all stipulations of this protocol, the conditions of IRB approval, 45 CFR Part 46, 21 CFR Part 50, 21 CFR Part 56, 21 CFR Part 812, ISO-14155, and International Conference on Harmonisation Good Clinical Practice (ICH GCP).

The protocol, informed consent form(s), recruitment materials, and all participant materials will be submitted to the Institutional Review Board (IRB) for review and approval. Approval of both the protocol and the consent form must be obtained before any participant is enrolled. Any amendment to the protocol will require review and approval by the IRB before the changes are implemented to the study. In addition, all changes to the consent form will be IRB-approved; a determination will be made regarding whether a new consent needs to be obtained from participants who provided consent, using a previously approved consent form.

#### 1. PURPOSE

The objective of this study is to compare the noninvasive hemoglobin (SpHb) performance of the Masimo Rainbow INVSENSOR00001 sensor against a control sensor. Data using the noninvasive devices will be collected from healthy volunteers undergoing a hemodilution procedure.

This is a nonrandomized single arm study wherein all subjects are enrolled into the experimental arm and receive both the INVSENSOR00001 sensor and the control sensor simultaneously on different fingers. Hemodilution will be conducted by delivery of intravenous fluids in a controlled manner to reduce the subject's blood concentration of hemoglobin to obtain noninvasive hemoglobin readings SpHb at various levels. Reference blood samples will be repeatedly collected from the subject and analyzed using a standard laboratory hematology analyzer. The performance of the sensors will be calculated using arithmetic root mean square (ARMS) analysis of the SpHb values and the reference blood values.

Outcome Measure: Comparison of INVSENSOR00001 and control SpHb sensor by ARMS calculation

Performance of the sensors will be determined by comparing the noninvasive hemoglobin measurement (SpHb) of the pulse oximeter sensors to the hemoglobin value obtained from a reference blood sample and calculating the ARMS value.

#### 2. BACKGROUND

Masimo Corporation develops non-invasive medical technologies. These devices have applications in the operating room, critical care unit, emergency room, emergency transport vehicles, as well as physician's offices.

A blood sample gives the best measure of hemoglobin as well as other blood solutes but is difficult to measure continuously and without skin puncture and risk of infection. Masimo SET and Masimo Rainbow technology allows real-time, non-invasive monitoring of hemoglobin (and other blood solutes) in patients and has the potential to improve clinical outcomes while reducing the cost of care and risks to both patients and clinicians associated with venipuncture.

#### 2.1. TECHNOLOGY BACKGROUND

Pulse oximetry is governed by the following principles:

- Oxyhemoglobin (oxygenated blood) and deoxyhemoglobin (non-oxygenated blood) differ in their absorption of red and infrared light (spectrophotometry).
- The amount of arterial blood in tissue changes with arterial pulses (photoplethysmography). Therefore, the amount of light absorbed by the varying quantities of arterial blood changes as well.

R-TP - 18788

# Comparison of Rainbow INVSENSOR00001 and Control SpHb Disposable Sensor Performance during Hemodilution

More generally, Masimo Pulse CO-Oximeters use a multi-wavelength sensor to distinguish between not only
oxygenated blood and deoxygenated blood, but also blood with carbon monoxide, oxidized blood and blood
plasma. The CO-Oximeter utilizes a sensor with various light-emitting diodes (LEDs) that pass light through
the site to a photodiode (detector). See figure below.



- Light Emitting Diodes (LEDs)
   (2+ wavelengths)
- 2. Detector
- Signal data is obtained by passing various visible and infrared lights through a capillary bed (for example, a
  fingertip, a hand, a foot) and measuring changes in light absorption during the blood pulsatile cycle. The
  detector receives the light, converts it into an electrical signal. Once the oximeter receives the signal from
  the sensor, it utilizes Masimo Rainbow signal extraction technology for calculation of the patient's
  hemoglobin level.

#### 2.2. STUDY DEVICES

Investigational sensor: INVSENSOR00001

The noninvasive, investigational INVSENSOR00001 sensor is a

The sensor has undergone risk assessment prior to use in human subjects to safeguard subject safety and well-being. Refer to the Investigator's Brochure for more details on the investigational device.

Control sensor: Masimo FDA-cleared SpHb disposable sensor

FDA-cleared Masimo Radical-7 pulse oximeter or equivalent

#### 3. REFERENCE

Consent Form

Post Care Instructions

Comparison of Rainbow INVSENSOR00001 and Control SpHb Disposable Sensor Performance during Hemodilution Case Report Form (CRF)

Comparison of Rainbow INVSENSOR00001 and Control SpHb Disposable Sensor Performance during Hemodilution Healthy Volunteers Needed Advertisement

Comparison of Rainbow INVSENSOR00001 and Control SpHb Disposable Sensor Performance during Hemodilution Recruitment Script

Comparison of Rainbow INVSENSOR00001 and Control SpHb Disposable Sensor Performance during Hemodilution Health Assessment Questionnaire

- Confidentiality Agreement

W-9 Request for Taxpayer Identification Number and Certification



R-TP - 18788

Comparison of Rainbow INVSENSOR00001 and Control SpHb Disposable Sensor Performance during Hemodilution



Volunteer payment form

#### 4. LOCATION

Masimo Corporation

Clinical Laboratory

52 Discovery

Irvine, CA 92618



#### 5. STUDY POPULATION

#### 5.1. Inclusion Criteria

- Competent adults between the ages of 18 and 50 years of age
- Must weigh a minimum of 110 lbs and no more than 250 lbs unless subject is over 6 feet tall
- BMI ≤ 35 unless the physician determines that a higher BMI is not due to morbid obesity, to safeguard subject safety during hemodilution
- Must have a hemoglobin value ≥ 11 g/dL at time of screening, , to safeguard subject safety during hemodilution
- Baseline heart rate between 45 bpm and 85 bpm
- CO value < 2.0% FCOHb
- Physical status of ASA I or II (American Society of Anesthesiology Class 1; Healthy subjects without
  any systemic disease at all. American Society of Anesthesiology Class II; subjects with mild systemic
  disease) The ASA definition strictly applies to the systemic disease portion of the classification
- Systolic BP ≤ 140 mmHg and Diastolic BP ≤ 90 mmHg
- Able to read and communicate in English

#### 5.2. Exclusion Criteria

- Pregnancy or positive hCG test
- Smokers (including e-cigarette users)
- Subject has known drug or alcohol abuse. Subjects who uses recreational drugs
- Subject has experienced a concussion or head injury with loss of consciousness within the last year
- Any chronic bleeding disorders (i.e. hemophilia)
- Any history of a stroke, myocardial infarction, or seizures
- Any cancer or history of cancer (not including skin cancer)

R-TP - 18788

# Comparison of Rainbow INVSENSOR00001 and Control SpHb Disposable Sensor Performance during Hemodilution



- Any cardiac dysrhythmias (i.e. atrial fibrillation)(without physicians clearance)
- Subject has known neurological and/or psychiatric disorder (i.e. schizophrenia, bipolar disorder) that interferes with the subject's level of consciousness
- Subject has Wolff-Parkinson-White Syndrome or Stokes-Adams Syndrome
- Subjects who have/are currently taking anticoagulant medication
- Subjects who have taken opioid pain medication within 24 hours of start of study
- Subjects who do not understand the study and the risks
- Subjects having either signs or history of peripheral ischemia
- Subjects who have had invasive surgery within the past year- including but not limited to major dental surgery, gallbladder, heart, appendix, major fracture repairs (involving plates/ screws), jaw surgery, urinary tract surgery, plastic surgery, major ENT surgery, joint replacement or gynecological surgeries, heart surgery or thoracic surgery
- Subjects that have symptoms of congestion, head colds, flu, or other illnesses
- Subjects with claustrophobia, or generalized anxiety disorder
- Subjects who have been in severe car accident(s) or a similar type of accident(s) requiring hospitalization within the last 12 months
- Subjects with chronic unresolved asthma, lung disease and respiratory disease
- Subjects with allergies to lidocaine, latex, adhesives, or plastic
- Subjects with heart conditions, insulin-dependent diabetes or uncontrolled hypertension
- Subjects who have given vaginal delivery, had a pregnancy terminated, a miscarriage with hospitalization or had a c-section within the last 6 months
- Subjects who intend on participating in any heavy lifting, repetitive movement of their wrist
  (including riding a motorcycle) or exercise (working out, riding a bike, riding a skate board etc.), or
  any activity that will put additional stress on the wrist within 24 hours following a study involving an
  arterial blood draw and/or arterial line placement
- Subject has any medical condition which in the judgment of the investigator and/or medical staff, renders them ineligible for participation in this study (Discretion of investigator)

#### 5.3. Withdrawal and replacement of subjects

Subjects must be withdrawn under the following circumstances:

- 5.3.1. The subject withdraws consent.
- 5.3.2. Discretion of investigator, for example: the investigator feels that the subject is too money motivated, the investigator feels that the subject does not fully comprehend and understand the consent form, the subject is ill-mannered and/or shows aggressive behavior towards study staff, malfunction of the device for greater than 30 minutes that prevents accurate collection of optical data.
- 5.4. Replacement of subjects

R-TP - 18788

# Comparison of Rainbow INVSENSOR00001 and Control SpHb Disposable Sensor Performance during Hemodilution



#### 6. EQUIPMENT AND MATERIALS

Equipment and Materials: All lab analyzers and equipment will be maintained per manufacturer specifications and all study personnel will be trained on the use of relevant equipment. Equivalent equipment and materials to those listed below may be used.

#### Subject safety monitoring equipment and medical supplies

- Non-invasive blood pressure arm cuff(s) as required
- ECG monitor FDA approved product
- Urine HCG pregnancy test
- Standard medical, wound care equipment and biohazard waste containers necessary to carry out the test procedure
- Standard Emergency equipment and medications will be available in the room during the study-Crash cart
- 0.5%-2% lidocaine as required
- Ethyl Chloride as required
- Pain Ease as required
- Heparin or saline flush solution (as required)- or equivalent



#### General lab supplies and equipment



#### 7. PROCEDURE

#### 7.1. SCHEDULE OF ACTIVITIES





R-TP - 18788

Masimo

Comparison of Rainbow INVSENSOR00001 and Control SpHb Disposable Sensor Performance during Hemodilution



#### 7.2. RECRUITMENT AND PRESCREENING

Subjects will be recruited using IRB-approved advertisements. Subjects may be referred to the study by previous volunteers. Subjects are contacted via phone call to conduct a prescreening interview to determine their initial eligibility for the study. Potential eligible subjects are scheduled for a study visit to the clinical laboratory.

#### 7.3. CONSENTING AND SCREENING

- 7.3.1. Study staff will discuss the informed consent process and the study with the potential subjects. The subjects will be provided with enough time to read and understand the informed consent document and their questions will be answered by study staff prior to the subject signing the informed consent form. No study related activities will be conducted until consent is signed.
- 7.3.2. The subject's weight and height are self-reported, however if the subject appears to be outside the weight range based on the inclusion/exclusion criteria, the subject will be weighed on a scale for verification.
- 7.3.3. Subjects will be asked to provide a copy of their valid government photo ID and/or Social Security card (SSN) to verify subject identity. The copies of these forms of identification will be stored along with the subject's consent. The confidentiality and retention of these documents will be protected to the extent provided and required by law.
- 7.3.4. Subjects will be asked a brief series of health questions to ensure their eligibility for this study. Subjects who do not meet the inclusion and exclusion criteria will not be eligible to participate in the study.



R-TP - 18788

Comparison of Rainbow INVSENSOR00001 and Control SpHb Disposable Sensor Performance during Hemodilution

- 7.3.5. Subject demographic information including age, sex, skin tone, ethnicity, height and weight will be collected. These may be recorded for data analysis and/or subject safety monitoring purposes.
- 7.3.6. In addition, a medical history will be recorded after the initial screening questionnaire.
- 7.3.7. Pre-procedure vital signs will be recorded for subject safety monitoring. Spikes in blood pressure and heart rate can be expected during line placement, needle sticks, blood draws etc. and may also be attributed to anxiety/nervousness relating to a new environment. Only the initial recorded blood pressure and/or heart rate determines a subject's qualification for the study.
- 7.3.8. Female subjects will be required to take a pregnancy test. Results will be noted in study documentation. If the pregnancy test is positive, the subject will be notified and removed from the study.
- 7.3.9. A venous sample will be obtained via needle stick or by placement of an IV and analyzed to verify that the subject meets the inclusion criteria for hemoglobin level. The subject will be excluded from the study if the values from the blood draw fall outside the ranges stated in the inclusion criteria.
- 7.3.10.
- 7.3.11. Subjects may be offered a snack (e.g., granola bar) and/or beverage (e.g., water, juice) due to the amount of time their involvement in this study may take.

#### 7.4. **PROCEDURES**

7.4.1. Standard hospital-type monitors will be placed on the subject, including ECG and blood pressure, for safety monitoring by medical staff. The procedure will be stopped if there is any evidence of volunteer stress or distress. These signs include but are not limited to a rise or fall in mean arterial blood pressure of more than 30% from baseline, a rise in heart rate to more than 130 BPM, complaints of feeling faint, chest discomfort, GI distress, urinary discomfort or feelings of a bloated bladder, or alternation of mental status. Blood samples are also monitored for hemoglobin and/or blood oxygenation levels for subject safety.



7.4.4. A-line) will be placed in the radial artery of the volunteer's wrist. The A-line is placed to facilitate continuous blood pressure measurement for subject safety monitoring, to enable repeated removal of blood aliquots for reference hemoglobin values, to allow for determination of arterial blood gases (ABG), Hgb, Hct, as well as other non-infectious blood solutes.

R-TP - 18788

Comparison of Rainbow INVSENSOR00001 and Control SpHb Disposable Sensor Performance during Hemodilution

be placed on the subject's fingers. sensors will be placed on the subject's fingers and connected to the data collection system. 7.4.6. Upon successful placement of the sensors and the volunteer's indication that they are comfortable, a baseline set of blood samples will be obtained. 7.4.8. Following removal of blood, the volunteer will rapidly receive intravenous fluid 7.4.11. The total amount of blood removed from the subject may be 7.4.13. Subjects may be warmed for their comfort 7.4.14. The hemodilution procedure will continue until the subject's fluid limits have been reached 7.4.15. The sensors/devices used in this study may be placed and removed by several operators multiple times during the study. 7.4.16. At the conclusion of the procedure, the sensors/devices, IV(s) and the arterial line(s) will be removed and the volunteer will be allowed to leave after medical personnel determine it is safe to do so.

7.4.18. All volunteers will be encouraged to remain in the study area until they feel fit to leave.

Subjects should feel safe and able before returning to work directly after participation in the

7.4.5. After arterial access is established, optical sensors for the noninvasive measurement(s) will

R-TP - 18788

# Comparison of Rainbow INVSENSOR00001 and Control SpHb Disposable Sensor Performance during Hemodilution

study. Subjects who are employees of Masimo will be advised to take as much time as they need after the study before returning to work.

- 7.4.19. Volunteers will be given instructions on wound care. All volunteers will be instructed to contact the principal investigator in the event of any potential complication.
- 7.4.20. The total time for the study procedures will be up to approximately event that the total procedure time exceeds subjects will be compensated for the extra time. Volunteers will be paid according to the compensation breakdown on the consent form.
- 7.4.21. Subjects will be provided with information related to any significant new findings that develop at any time during the study which may relate to their willingness to continue their participation, their health and/or medical care.

#### 8. ACCEPTANCE CRITERIA

The sensors will be determined to have equivalent performance based on the agreement of their ARMS values.

#### 9. SAMPLE SIZE JUSTIFICATION AND DATA ANALYSIS PROCEDURE TO BE USED

9.1. Sample size determination

Sample size for this study has been determined to be based on previous experience with similar devices and Masimo internal procedures for sample size calculation and justification

9.2. Statistical Analysis

Accuracy will be reported as the A<sub>RMS</sub> using the following equation:

$$Bias = \frac{1}{n} \sum_{i=1}^{n} (SpHb - tHb)$$

$$Precision = \sqrt{\frac{\sum_{i=1}^{n} ((SpHb - tHb) - Bias)^{2}}{n}}$$

$$A_{RMS} = \sqrt{\frac{\sum_{i=1}^{n} (SpHb - tHb)^{2}}{n}}$$

9.3. Measures taken to minimize/avoid bias:

9.3.2. Operators will not make any decisions based on results from other operators or any parameters obtained from blood samples.

9.4. Expected drop out rates

Subjects may not complete the study for various reasons, such as screen failure, unable to complete hemodilution criteria, unable to have intravenous or arterial line placed.



R-TP - 18788

Comparison of Rainbow INVSENSOR00001 and Control SpHb Disposable Sensor Performance during Hemodilution

#### 10. ADVERSE EVENTS

Definitions:

<u>Adverse event</u>: Any untoward medical occurrence in a subjects, users or other persons, whether or not related to the medical device under study.

<u>Device-related adverse event</u>: Adverse event related to, associated with, or caused by, the use of a medical device under study, including but not limited to events that may have been attributed to the device because of device failure or malfunction, improper or inadequate design, manufacture or user error.

<u>Device deficiency</u>: Inadequacy of a medical device with respect to its identity, quality, durability, reliability, safety or performance. Device deficiencies include malfunctions, use errors and inadequate labeling.

<u>Serious adverse event</u>: Adverse event that: a) led to death, b) led to serious deterioration in the health of the subject, that resulted in: (i) a life-threatening illness or injury, (ii) a persistent or significant impairment of a body structure or a body function, (iii) in-patient or prolonged hospitalization, or (iv) medical or surgical intervention to prevent life-threatening illness or injury or permanent impairment to a body structure or a body function, or c) led to fetal distress, fetal death or a congenital abnormality or birth defect. NOTE: Planned hospitalization for a pre-existing condition, or a procedure required by the clinical investigational plan, without serious deterioration in health, is not considered a serious adverse event.

All adverse events will be reported and documented as described below.

#### 10.1. Adverse Events

All adverse events that occur during the study shall be recorded on the Case Report Form even if the investigator assesses the adverse event as unlikely to be causally related to the test device or study procedures. The investigator will inform the sponsor and IRB as required by IRB reporting guidelines.

#### 10.2. Serious Adverse Events

- 10.2.1 The investigator/study staff shall promptly report both serious adverse events (e.g., subject death, subject hospitalization for several days) and unanticipated adverse device effects to the sponsor within 48 hours. All serious adverse events will also be reported to the IRB per IRB reporting requirements.
- 10.2.2 At the time of discharge from the study, any unresolved serious adverse event(s) will be followed up by the investigator until the event(s) are resolved, stabilized or the patient is lost to follow-up or the adverse event is otherwise explained. The investigator will also instruct the subject to report any subsequent events occurring in the next 30 days, which the subject or the subject's physician believes might reasonably be regarded as caused by or have a reasonable possibility of being caused by the test device or procedures involved in the study.

#### 10.3. Unanticipated Problems

Any unanticipated problem involving subjects or others will be reported to the IRB, such as protocol violations or deviations as required by the IRB reporting procedures.

#### 11. SUPPORTING DOCUMENTATION AND OPERATIONAL CONSIDERATIONS

- 11.1. Measures Taken to Protect the Rights and Welfare of Subjects
  - 11.1.1. All subjects will be monitored closely throughout the study. There will be an ACLS certified medical doctor present in the study area throughout the study.

R-TP - 18788

# Comparison of Rainbow INVSENSOR00001 and Control SpHb Disposable Sensor Performance during Hemodilution

- 11.1.2. The following measures will be taken to ensure the confidentiality of the subjects:
  - 11.1.2.1.A code (identification) number for each subject will be kept on file.
  - 11.1.2.2.Only their corresponding identification number will identify subjects.
  - 11.1.2.3. Access to identifying documents (IC, SSN, photo ID) and data will only be made to the principal investigators in the study and study staff.
  - 11.1.2.4. The confidentiality and retention of these documents will be protected to the extent provided and required by the law.

#### 11.2. Vulnerable Populations

11.2.1. Employees are considered to be a vulnerable population.

Participation is not a condition of employment. There will be no repercussions in the workplace in the case that the employee refuses to participate in the study or withdraws at any point during the study. Neither supervisors nor superiors will be involved in the recruitment of employees for participation in the study.

11.2.2. Economically disadvantaged or unemployed and educationally disadvantaged

Reasonable compensation will be provided for economically disadvantaged subjects to eliminate possibility of undue influence due to financial incentive. Educationally disadvantaged subjects will be provided ample time to ask questions and comprehend information.

#### 11.3 Documents and Database

| made. If destroyed, these documents will | be shredded and done by a certified company used for |
|---|---|
| destroying medical and clinical data | |

#### 12. DEVICE ACCOUNTABILITY

#### 12.1. Receipt of Study Device

Upon receipt of the study device supplies, an inventory must be performed and the device accountability log filled out and signed by the person accepting the shipment. It is important that the designated study staff counts and verifies that the shipment contains all the items noted in the shipment inventory. Any damaged or unusable study devices in a given shipment will be documented in the study files.

12.2. Use of Study Device

Use of devices and sensors will be documented on case report forms for each subject.



R-TP - 18788

# Comparison of Rainbow INVSENSOR00001 and Control SpHb Disposable Sensor Performance during Hemodilution

12.3. Return or Destruction of Study Device

At the completion of the study, there will be a final reconciliation of study devices and sensors shipped, devices/sensors used, and devices/sensors remaining. This reconciliation will be logged on the device accountability log. Any discrepancies noted will be investigated, resolved, and documented prior to return or destruction of unused study devices. Devices destroyed on site will only be upon written instruction from the sponsor and will be documented in the study files.

#### 13. RISKS AND BENEFITS

- 13.1. Benefits: There would be no other benefit to the subject. Other possible benefits would be to society as a whole. Evaluation of the accuracy of this new device could enable healthcare workers to more appropriately treat potentially life threatening conditions.
- 13.2. Device Risks: The noninvasive devices used in this study are similar in technology and design to some commercially available pulse oximeters and other non-invasive devices and hence have the same risks. Pulse oximeters and other non-invasive devices are commonly used and are considered to be minimal risk. There is an extremely small risk of damage to the subject's fingers, or other locations where sensors are placed, from the device including temporary skin irritation or discomfort associated with exposure to the sensor as well as potential temporary mechanical irritation or discomfort. There is a remote, yet possible, risk of a burn from the sensor. In the case of a sensor burn there is the potential for permanent skin damage (scar/discoloration).
- 13.4. Arterial Cannulation risks: bleeding, infection, hematoma, damage to the blood vessel and surrounding nerves, tendons or tissue; loss of feeling in hand and/or arm and even the loss of hand due to rare complications of the study.
- 13.5. Risks Associated with Removal of Blood: Removal of blood is generally considered to be safe in most patients and exceptionally safe in healthy volunteers (i.e. blood donation). The risk of removing blood includes the risks obtaining venous access. Additionally, there is the risk of hypotension, tachycardia, anemia, dizziness and loss of consciousness. All subjects will be maintained in a reclined position throughout the study and a physician will be available to continually monitor the vital signs.
- 13.6. Blood Draw risks: discomfort is generally associated with needle puncture. The most common complications associated with blood draws and capillary sticks are hematomas or bruising. All blood draws will be performed by qualified personnel. An ACLS certified physician will be in attendance throughout the entire procedure, and the study will be completed under their general supervision. Other anticipated adverse events that may occur, include but are not limited to: Vaso vagal (passing out), infiltrated IV, lightheadedness, feeling flush/ warm, feeling nauseated, throwing up, seizures, sudden drop in blood pressure/ sudden increase in blood pressure, sudden drop in heart rate/ sudden increase in heart rate, tingling sensation of face/arms and/or sweating, and mouth dryness. These anticipated adverse events are expected to be temporary.
- 13.7. Risk From Hemodilution: Hemodilution has been used successfully as a technique to reduce perioperative blood loss during surgery. Hemodilution is generally considered to be safe in most patients and exceptionally safe in healthy volunteers. In surgery, the chief benefit of hemodilution is the reduction of blood losses when whole blood is shed perioperatively at lower hematocrit levels after hemodilution is completed. In our controlled clinical lab, withdrawal and blood loss will be limited to samples required for laboratory analysis; hemodilution will be used principally to lower



R-TP - 18788

Comparison of Rainbow INVSENSOR00001 and Control SpHb Disposable Sensor Performance during Hemodilution

the subject's hematocrit and hemoglobin. The risks of hemodilution include heart failure, respiratory failure, hypertension, edema, infection and electrolyte abnormalities. Isotonic fluids will be administered. A physician will be immediately available thorough out the procedure and vital signs will be continually monitored.



- 13.10. Risk From Loss of Confidentiality: Masimo upholds the highest standards to protect hard and electronic data however a complete promise for confidentiality cannot be guaranteed due to unforeseeable events.
- 13.11. Risk From Additional Testing:

will refer them to their primary care physician.

- 13.11.1.During the conduct of the study, it is possible, but not likely, that someone could become exposed to the sample of blood drawn from the subject through an inadvertent needle stick or by contact with an open cut. In such circumstances, it will be important to the exposed individual to know whether the blood to which he or she was exposed contained Hepatitis B virus (HBV), Human immunodeficiency virus (HIV), or Hepatitis C virus (HCV) and additional testing of the sample will be performed.
- 13.11.2.Within the consent subjects will agree to permit the company to test the blood sample (or samples) by signing the consent. The test results will be maintained as confidential and will only be used by healthcare professionals for the diagnosis and treatment of the exposed individual as appropriate.
- 13.11.3.In the case that Masimo needs to contact a subject regarding additional testing they will be contacted by a Masimo employee and medical personnel can be available for further counsel if requested.
- 13.11.4. The cost for the initial testing and compensation for their time/travel to the testing facility will be the only things paid for by Masimo.
- 13.12. Lidocaine (injection) Risks: Insertion of the Lidocaine may be discomforting and can feel like a slight pinch along with a warm/burning sensation. Other anticipated adverse events that may occur, include but are not limited to: Flushing or redness of the skin, itching skin, small red or purple spots on the skin, unusually warm skin, bruising, bleeding at the application site, swelling. These adverse events are expected to be temporary.
- 13.13. Although not common, it is also possible to have an allergic reaction to injectable lidocaine. Subjects should not take part in this study if they are allergic to lidocaine injection or other types of numbing medicine, or if they have a heart rhythm disorder such as Wolff-Parkinson-White Syndrome or



R-TP - 18788

# Comparison of Rainbow INVSENSOR00001 and Control SpHb Disposable Sensor Performance during Hemodilution



13.14. Ethyl Chloride (Lidocaine Spray): Ethyl Chloride is a topical anesthetic which is used to prevent pain by cooling the skin. Although unlikely, the anticipated adverse events that may occur, include but are not limited to: changes in skin color (i.e. Flushing or redness of the skin), delayed wound healing, rash, itching and swelling. These adverse events are expected to be temporary.

#### 14. EMERGENCY RESPONSE PLAN FOR MEDICAL EMERGENCIES

The physician and nurse present during the study will be ACLS certified and will respond to any medical emergency involving a volunteer with the ACLS approved protocol for intervention. A crash cart is on site and full emergency services are within 3 miles.

#### 15. MONITORING PLAN

A separate document for the study monitoring plan will be developed and followed to ensure subject safety and GCP compliance.

#### 16. PROTOCOL DEVIATIONS AND AMENDMENTS

Deviations to the protocol will be documented on the Case Report Form or a separate document. Protocol deviations will be reported to the sponsor and IRB per IRB reporting guidelines.

Modifications to the protocol, informed consent materials, recruitment materials, or any other materials provided to subjects must be reviewed and approved by the IRB.